CLINICAL TRIAL: NCT05762991
Title: Application of Artificial Intelligence on the Diagnosis of Helicobacter Pylori Infection and Premalignant Gastric Lesion: A Multihospital Study
Brief Title: Application of Artificial Intelligence on the Diagnosis of Helicobacter Pylori Infection and Premalignant Gastric Lesion
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202111108RINC
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Helicobacter Pylori Infection; Premalignant Lesion
Keywords: Helicobacter, Artificial Intelligence, Telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Helicobacter pylori infection and premalignant gastric lesion: Application of artificial intelligence to analyze the correlation between endoscopic images and urea breath test results/histopathological results.

SUMMARY:
The aim of this diagnostic accuracy study is to evaluate the application of artificial intelligence on the diagnosis of Helicobacter pylori infection and premalignant gastric lesions based on upper endoscopic images. We use techniques of artificial intelligence to analyze the correlation between endoscopic images and urea breath test results/histopathological results.

DETAILED DESCRIPTION:
This study had invited patients to undergo urea breath test, upper gastrointestinal endoscopy, and histology examination. The study will collect their tests results, upper gastrointestinal endoscopy images, and histopathological results. Artificial intelligence techniques will be used to analyze the correlation between endoscopic images and urea breath test results/histopathological results. We aim to establish a telemedicine system to assist clinicians in diagnosing Helicobacter pylori infection and detecting premalignant gastric lesion using upper endoscopic images. The system will be implemented as a telemedicine service system in the rural areas, for example Matsu Islands. The baseline histological predictions will be linked to the newly incident gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-80
2. Scheduled urea breath test and endoscopy

Exclusion Criteria:

1. History of gastric surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will invite patients who need to undergo urea breath test, upper gastrointestinal endoscopy and histology examination.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity to detect premalignant gastric lesions | Up to 5 years
  Outcomes include the atrophic gastritis, intestinal metaplasia, and Helicobacter pylori infection

SECONDARY OUTCOMES:
Specificity to exclude premalignant gastric conditions | Up to 5 years
  Outcomes include the atrophic gastritis, intestinal metaplasia, and Helicobacter pylori infection

OTHER OUTCOMES:
Areas under the ROC curves | Up to 5 years
  Outcomes include the atrophic gastritis, intestinal metaplasia, and Helicobacter pylori infection
Gastric cancer incidence | Up to 10 years
  New incident gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hsien Chiang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Yi-Chia Lee, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The study was based on the images and histological data.